CLINICAL TRIAL: NCT00937664
Title: A Phase I, Open-Label, Dose-Escalation Study to Assess Safety, Tolerability & Pharmacokinetics of AZD7762 Administered as a Single Intravenous Agent and in Combination w/ Wkly Standard Dose Gemcitabine in Japanese Patients w/ Advanced Solid Malignancies
Brief Title: Safety and Tolerability Study of AZD7762 in Combination With Gemcitabine
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Termination of the study was made after a full review of program data and assessment of the current risk-benefit profile.
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1040C00008
Record Dates: First submitted 2009-07-09; First posted 2009-07-13 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Cancer; Solid Tumors; Advanced Solid Malignancies
Keywords: Phase I; cancer; solid tumors; advanced solid malignancies; dose escalation; combination treatment; CHK inhibitor; Japanese
MeSH Terms: conditions — Neoplasms | interventions — 3-(carbamoylamino)-5-(3-fluorophenyl)-N-(3-piperidyl)thiophene-2-carboxamide; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD7762 + gemcitabine (Other): AZD7762 administered alone and in combination with gemcitabine
  Interventions: Drug: AZD7762; Drug: gemcitabine

INTERVENTIONS:
Drug: AZD7762 — solution, intravenous, weekly
Drug: gemcitabine — intravenous, weekly
  Other Names: Gemzar

SUMMARY:
The primary purpose of this study is to find out what the maximum tolerated dose is for an experimental drug called AZD7762 when given with the approved drug gemcitabine based on the side effects experienced by patients that receive both drugs.

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients with advanced solid tumors for which standard treatment does not exist or is no longer effective.
* Must be suitable for treatment with gemcitabine
* Relatively good overall health other than cancer

Exclusion Criteria:

* Poor bone marrow function (not producing enough blood cells).
* Poor liver or kidney function.
* Serious heart conditions

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of adverse events (based on CTCAE version 3.0), laboratory values, vital sign measurements, cardiac markers, ECG, Echocardiogram | Laboratory values weekly for all treatment cycles, and the other variables weekly for Cycle 0-1, then every cycle (3-4 weeks) from Cycle 2

SECONDARY OUTCOMES:
Pharmacokinetic effect of AZD7762 when administered alone and in combination with gemcitabine | According to protocol specified schedule, the number of PK samples collected during Cycle 0 and Cycle 1
Anti-tumor activity of AZD7762 when administered in combination with gemcitabine by assessment of Response Evaluation Criteria in Solid Tumors (RECIST) | Every 2-3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Peter Langmuir, MD, Study Director — AstraZeneca; Takashi Seto, MD, PhD, Principal Investigator — National Hospital Organization Kyushu Cancer Center
Locations (1):
- Research Site, Minamiku, Fukuoka, Japan